CLINICAL TRIAL: NCT02791334
Title: A Phase 1a/1b Study of a Novel Anti-PD-L1 Checkpoint Antibody (LY3300054) Administered Alone or in Combination With Other Agents in Advanced Refractory Solid Tumors (Phase 1a/1b Anti-PD-L1 Combinations in Tumors-PACT)
Brief Title: A Study of Anti-PD-L1 Checkpoint Antibody (LY3300054) Alone and in Combination in Participants With Advanced Refractory Solid Tumors
Acronym: PACT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16088; I8J-MC-JYCA (Other: Eli Lilly and Company); 2016-000440-33 (EudraCT Number)
Record Dates: First submitted 2016-06-01; First posted 2016-06-06 (Estimated); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Solid Tumor; Microsatellite Instability-High (MSI-H) Solid Tumors; Cutaneous Melanoma; Pancreatic Cancer; Breast Cancer (HR+HER2-)
Keywords: PDL1; PD-L1
MeSH Terms: conditions — Melanoma; Pancreatic Neoplasms; Breast Neoplasms | interventions — LY3300054; Ramucirumab; abemaciclib; merestinib; LY3321367

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- LY3300054 (Experimental): LY3300054 given intravenously (IV) on day 1 and day 15 of a 28 day cycle or LY3300054 given IV on day 1 of a 21 (or 28) day cycle.
  Interventions: Drug: LY3300054
- LY3300054 + Ramucirumab (Experimental): LY3300054 and ramucirumab given IV on day 1 and day 15 of a 28 day cycle or ramucirumab given IV on day 1 and day 8 and LY3300054 given IV on day 1 of a 21 day cycle.
  Interventions: Drug: LY3300054; Drug: Ramucirumab
- Abemaciclib + LY3300054 (Experimental): LY3300054 given IV on day 1 and day 15 and abemaciclib given orally every 12 hours of a 28 day cycle.
  Interventions: Drug: LY3300054; Drug: Abemaciclib
- LY3300054 + Abemaciclib (Concurrent Dosing) (Experimental): LY3300054 given IV on day 1 and day 15 and abemaciclib given orally every 12 hours of a 28 day cycle.
  Interventions: Drug: LY3300054; Drug: Abemaciclib
- LY3300054 + Abemaciclib (Experimental): LY3300054 given IV on day 1 and day 15 and abemaciclib given orally every 12 hours of a 28 day cycle. This arm will only be initiated if required.
  Interventions: Drug: LY3300054; Drug: Abemaciclib
- LY3300054 + Merestinib (Experimental): LY3300054 given IV on day 1 and day 15 and merestinib given orally once daily of a 28 day cycle.
  Interventions: Drug: LY3300054; Drug: Merestinib
- LY3300054 Expansion (Metastatic Cutaneous Melanoma) (Experimental): LY3300054 given IV on day 1 and day 15 of a 28 day cycle.
  Interventions: Drug: LY3300054
- LY3300054 Expansion (MSI-H Solid Tumors) (Experimental): LY3300054 given IV on day 1 and day 15 of a 28 day cycle.
  Interventions: Drug: LY3300054
- : LY3300054 + Abemaciclib (HR+, HER2- Breast Cancer) Expansion (Experimental): LY3300054 given IV on day 1 and day 15 and abemaciclib given orally every 12 hours of a 28 day cycle.
  Interventions: Drug: LY3300054; Drug: Abemaciclib
- LY3300054 + LY3321367 Expansion (PD-1/PD-L1 Naïve, MSI-H) (Experimental): LY3300054 and LY3321367 given IV on day 1 and day 15 of a 28 day cycle.
  Interventions: Drug: LY3300054; Drug: LY3321367
- LY3300054 + LY3321367 Expansion (Experimental): LY3300054 and LY3321367 given IV on day 1 and day 15 of a 28 day cycle.
  Interventions: Drug: LY3300054; Drug: LY3321367
- LY3300054 + Merestinib (Pancreatic Cancer) Expansion (Experimental): LY3300054 given IV on day 1 and day 15 and merestinib given orally once daily of a 28 day cycle.
  Interventions: Drug: LY3300054; Drug: Merestinib

INTERVENTIONS:
Drug: LY3300054 — Administered IV
Drug: Ramucirumab — Administered IV
  Other Names: LY3009806
  Arms: LY3300054 + Ramucirumab
Drug: Abemaciclib — Administered orally
  Other Names: LY2835219
  Arms: : LY3300054 + Abemaciclib (HR+, HER2- Breast Cancer) Expansion; Abemaciclib + LY3300054; LY3300054 + Abemaciclib; LY3300054 + Abemaciclib (Concurrent Dosing)
Drug: Merestinib — Administered orally
  Other Names: LY2801653
  Arms: LY3300054 + Merestinib; LY3300054 + Merestinib (Pancreatic Cancer) Expansion
Drug: LY3321367 — Administered IV
  Arms: LY3300054 + LY3321367 Expansion; LY3300054 + LY3321367 Expansion (PD-1/PD-L1 Naïve, MSI-H)

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of anti-programmed cell death ligand 1 (PD-L1) checkpoint antibody LY3300054 in participants with advanced refractory solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic confirmation of advanced solid tumor.
* For LY3300054 + abemaciclib only: No participants with liver metastases. Participants must have normal aspartate aminotransferase (AST), alanine aminotransferase (ALT), total bilirubin, direct bilirubin.
* For LY3300054 + abemaciclib in HR+, HER- breast cancer:

  * Express at least 1 of the hormone receptors [HR; estrogen receptor (ER) or progesterone receptor (PR)] by immunohistochemistry (IHC) to fulfill the requirement for HR+ disease on the primary tumor or metastatic lesion of the breast cancer. ER and PR assays are considered positive if there is at least 1% positive tumor nuclei in their sample as defined in the relevant American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) or local guidelines.
  * To fulfill the requirement of HER2- disease, a breast cancer must not demonstrate, at initial diagnosis or upon subsequent biopsy, overexpression of HER2 by either IHC or in-situ hybridization (ISH) as defined in the relevant ASCO/CAP or local guidelines.
  * Most recent HR and HER2 receptor testing should be used to determine eligibility.
  * Have previously received prior treatment with at least 1 but no more than 3 chemotherapy regimens in the metastatic setting.
  * Have AST, ALT, GGT, and AP that are ≤2.5x upper limit of normal (ULN) and normal bilirubin (total and direct) regardless of liver involvement.
* For LY3300054 + merestinib in pancreatic cancer:

  * Histologically or cytological confirmed diagnosis of metastatic or locally advanced, unresectable pancreatic adenocarcinoma (excluding other pancreatic malignancies for example, acinar cell carcinomas, adenosquamous carcinomas, and neuroendocrine islet cell neoplasms).
  * Have had disease progression, be refractory or intolerant to no more than 2 prior systemic regimens.
* For LY3300054 + LY3321367 in PD-1/PD-L1-naive, MSI-H/MMR-deficient advanced solid tumors:

  * Have histologically or cytologically confirmed diagnosis of advanced solid tumor AND shown to be MSI-H or MMR-deficient.
* For LY3300054 + LY3321367 in PD-1/PD-L1- resistant/refractory, MSI-H/MMR-deficient advanced solid tumors:

  * Have histologically or cytologically confirmed diagnosis of advanced solid tumor AND shown to be MSI-H or MMR-deficient.
  * Prior exposure to PD-1/PD-L1 agent regardless of response.
* For Phase 1b LY3300054 monotherapy or combination therapy, no prior treatment with a PD-1 or PD-L1 agent is allowed.

  * Exception: the LY3321367 combination in participants with PD-1/PD-L1- resistant/refractory, MSI-H, where prior exposure to PD-1/PD-L1 agent required.
* For Phase 1a LY3300054 monotherapy or combination therapy, previous immunotherapy is acceptable if the following criteria are met:

  * Must not have experienced a toxicity that led to permanent discontinuation of prior immunotherapy.
  * Must have completely recovered or recovered to baseline prior to screening from any prior adverse events (AEs) occurring while receiving prior immunotherapy.
  * Must not have experienced a Grade ≥3 immune-related AE or an immune-related neurologic or ocular AE of any grade while receiving prior immunotherapy.
  * Must not have required the use of additional immunosuppressive agents other than corticosteroids for the management of an AE, not have experienced recurrence of an AE if re-challenged, and not currently require maintenance doses of >10 milligrams prednisone or equivalent per day.
* Have at least 1 measurable lesion assessable using standard techniques by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
* Have adequate organ function.
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) scale.
* Have an estimated life expectancy of ≥12 weeks, in the judgment of the investigator.
* Have submitted a tumor tissue sample, as follows:

  * For participants entering the Phase 1a dose escalation: have submitted, if available, the most recent archival tumor tissue sample.
  * For those participating ONLY in Phase 1b expansions: Have submitted tumor tissue sample from a newly obtained core or excisional biopsy for a tumor lesion (preferred) or a recent biopsy taken with 3 months prior to study enrollment and following the participants most recent prior systemic treatment and be willing to undergo a biopsy procedure during the study treatment period for collection of additional tumor tissue sample.

Exclusion Criteria:

* Have a serious concomitant systemic disorder including human immunodeficiency virus (HIV), active hepatitis B virus (HBV), active hepatitis C virus (HCV), active autoimmune disorder or disease requiring high dose of steroids.
* Have a bowel obstruction, history or presence of inflammatory enteropathy or extensive intestinal resection or chronic diarrhea.
* Have evidence of interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity or active, noninfectious pneumonitis.
* Have an active infection requiring systemic therapy.
* Have moderate or severe cardiovascular disease.
* Have symptomatic or uncontrolled brain metastases, spinal cord compression, or leptomeningeal disease requiring concurrent treatment.
* Have received a live vaccine within 30 days before the first dose of study treatment.
* Have a significant bleeding disorder or vasculitis or had a Grade ≥3 bleeding episode within 12 weeks prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2016-06-29 (Actual); Primary Completion 2020-05-22 (Actual); Study Completion 2024-06-27 (Actual)

PRIMARY OUTCOMES:
Number of Participants with LY3300054 Dose Limiting Toxicities (DLTs) | Baseline through Cycle 1 (Approximately 28 Days)

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY3300054 | Predose Cycle 1 Day 1 Through Follow Up (Approximately 6 Months)
PK: Cmax of Ramucirumab | Predose Cycle 1 Day 1 Through Follow Up (Approximately 6 Months)
PK: Cmax of Abemaciclib | Predose Cycle 1 Day 1 Through Follow Up (Approximately 6 Months)
PK: Cmax of Merestinib | Predose Cycle 1 Day 1 Through Follow Up (Approximately 6 Months)
PK: Cmax of LY3321367 | Predose Cycle 1 Day 1 Through Follow Up (Approximately 6 Months)
Objective Response Rate (ORR): Proportion of Participants With a Complete Response (CR) or Partial Response (PR) | Baseline to Measured Progressive Disease (Approximately 6 Months )
Progression Free Survival (PFS) | Baseline to Measured Progressive Disease or Death (Approximately 12 Months)
Duration of Response (DoR) | Date of CR or PR to Date of Measured Progressive Disease or Death Due to Any Cause (Approximately 12 Months)
Time to Response (TTR) | Baseline to Date of CR or PR (Approximately 6 Months)
Disease Control Rate (DCR): Proportion of Participants who Exhibit Stable Disease (SD), CR or PR | Baseline to Measured Progressive Disease (Approximately 6 Months)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (14):
- United States (3):
  - Tennessee Oncology PLLC, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - The START Center for Cancer Care, San Antonio, Texas
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
- Princess Margaret Hospital, Toronto, Ontario, Canada
- France (2):
  - Institut Bergonié - Centre Régional de Lutte Contre Le Cancer de Bordeaux et Sud Ouest, Bordeaux
  - Gustave Roussy, Villejuif
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
- Spain (2):
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Madrid Norte Sanchinarro, Madrid
- Taiwan (2):
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei

REFERENCES:
- [Derived] Hollebecque A, Chung HC, de Miguel MJ, Italiano A, Machiels JP, Lin CC, Dhani NC, Peeters M, Moreno V, Su WC, Chow KH, Galvao VR, Carlsen M, Yu D, Szpurka AM, Zhao Y, Schmidt SL, Gandhi L, Xu X, Bang YJ. Safety and Antitumor Activity of alpha-PD-L1 Antibody as Monotherapy or in Combination with alpha-TIM-3 Antibody in Patients with Microsatellite Instability-High/Mismatch Repair-Deficient Tumors. Clin Cancer Res. 2021 Dec 1;27(23):6393-6404. doi: 10.1158/1078-0432.CCR-21-0261. Epub 2021 Aug 31. PMID 34465599
- [Derived] Patnaik A, Yap TA, Chung HC, de Miguel MJ, Bang YJ, Lin CC, Su WC, Italiano A, Chow KH, Szpurka AM, Yu D, Zhao Y, Carlsen M, Schmidt S, Vangerow B, Gandhi L, Xu X, Bendell J. Safety and Clinical Activity of a New Anti-PD-L1 Antibody as Monotherapy or Combined with Targeted Therapy in Advanced Solid Tumors: The PACT Phase Ia/Ib Trial. Clin Cancer Res. 2021 Mar 1;27(5):1267-1277. doi: 10.1158/1078-0432.CCR-20-2821. Epub 2020 Nov 23. PMID 33229456
- See also: A Study of Anti-PD-L1 Checkpoint Antibody (LY3300054) Alone and in Combination in Participants With Advanced Refractory Solid Tumors — https://trials.lillytrialguide.com/en-US/trial/3RHxoNIFMkcEKKcQe8uMCW